

# Multicenter Prospective Randomized Control Study on Persona Total Knee System vs NexGen Total Knee System in Total Knee Arthroplasty

#### K.CR.I.EU.15.13

Protocol no.: 1.05

November 28th, 2016

#### **Primary investigator**

Anders Troelsen, MD, Professor. (1) (Surgeon)

Kirill Gromov, MD (1) (Surgeon)

## **Investigators**

Henrik Husted, MD (1) (Surgeon)

Per Wagner Kristensen, MD (2) (Surgeon)

Andreas Kappel, MD (3) (Surgeon)

Henrik Schrøder, MD (4) (Surgeon)

Anders Odgaard, MD (5) (Surgeon)

# **Sponsor**

Zimmer Biomet



## **Investigating institutions in Denmark**

1) Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre (1)

DK-2650 Hvidovre, Copenhagen, Denmark

2) Dept. of Orthopaedic Surgery, Vejle Sygehus, Sygehus Lillebælt (3)

DK-7100, Vejle, Denmark

3) Dept. of Orthopaedic Surgery, Farsø Sygehus, Ålborg Universitetshospital (4)

DK-9000, Aalborg, Denmark

4) Dept. of Orthopaedic Surgery, Næstved Sygehus, (5)

DK-4700, Næstved, Denmark

5) Dept. of Orthopaedic Surgery, Copenhagen University Hospital Gentofte, (6)

DK-2900, Hellerup, Denmark

#### Institution for radiographic data analysis and data collection

1) Dept. of Orthopaedic Surgery, Copenhagen University Hospital Hvidovre (1)

DK-2650 Hvidovre, Copenhagen, Denmark.



# **Study Synopsis**

| TITLE | Multicenter Prospective Randomized Control Study on Persona Total Knee System vs<br>NexGen Total Knee System in Total Knee Arthroplasty |
|---|---|
| PROTOCOL NUMBER | K.CR.I.EU.15.13 (RCT) |
| STUDY DESIGN | Multicenter, 2-arm, randomized, controlled, single-blinded post-market study |
| STUDY OBJECTIVES /<br>ENDPOINTS | <ul> <li>Multicenter, 2-arm, randomized, controlled, single-blinded post-market study</li> <li>Primary endpoint: <ul> <li>Evaluate patient reported outcome measures following primary total knee replacement using Persona Total Knee system compared to NexGen total Knee System as measured by: Oxford Knee Score (3 months, 1 and 2 years postoperatively)</li> </ul> </li> <li>Secondary endpoints: <ul> <li>Evaluate patient reported outcome measures following primary total knee replacement using Persona Total Knee system compared to NexGen total Knee System as measured by: Oxford Knee Score -Activity &amp; Participation Questionnaire (APQ) anchoring questions, EQ-5D and Forgotten Joint Score (3 months, 1 and 2 years postoperatively).</li> <li>Evaluate intra-operative and postop complications as well as long-term survivorship following primary total knee replacement using Persona Total Knee system compared to NexGen total Knee System as follows:</li></ul></li></ul> |
| | <ul> <li>Survival through registries at 5,7 and 10 years postoperatively.</li> </ul> |
| INCLUSION/EXCLUSION<br>CRITERIA | <ul> <li>Inclusion criteria: <ul> <li>Patients with clinical and radiological osteoarthritis of the knee set to receive a primary unilateral total knee replacement</li> <li>&gt;18 years of age</li> <li>Participants must be able to speak and understand Danish, able to give informed consent and be cognitively intact, able to complete all post-operative controls</li> <li>Participants must not have severe comorbidities, ASA score ≤ 3</li> <li>Patients should be clinically suitable to receive a CR implant (no severe deformity and/or ligament instability)</li> </ul> </li> <li>Exclusion criteria: <ul> <li>Terminal illness</li> <li>Revision knee replacement surgery</li> </ul> </li> </ul> |



| | <ul> <li>RA</li> <li>Traumatic etiology</li> <li>Prior surgery on the affected knee that includes osteosynthesis, ACL and/or PCL and/or collateral ligament surgery. Arthroscopy with menisceotomy / cartilage surgery / house cleaning is allowed.</li> <li>Altered pain perception and / or neurologic affection due to diabetes or other disorders.</li> <li>Patients will be excluded intraoperative if CR implant is not suitable</li> </ul> |
|---|---|
| SAMPLE SIZE | 314 patients |
| LENGTH OF STUDY | Start/End-date: 2016 / 2029 (18 months enrolment, 2 years postoperative visits, up to 10 years postoperative follow-up in the registries) |
| INVESTIGATIONAL PRODUCTS | <ul> <li>Persona Total Knee System</li> <li>NexGen total Knee System</li> <li>Only cruciate retaining (CR) components will be used in this study.</li> <li>Both cemented and cementless femoral components</li> <li>Both standard as well as narrow femoral components</li> <li>Only cemented tibial components</li> <li>Conventional polyethylene will be used for patients &gt;65 years old and Vitamin-E infused poly insert may be used for patients ≤ 65 years old.</li> <li>Resurfacing of patella is performed in all cases.</li> </ul> |
| SCORES/PERFORMANCE<br>ASSESSMENTS | OKS, OKS-APQ, EQ-5D, FJS, Patient satisfaction, ROM, X-rays (AP/lateral) |
| STATISTICAL REPORTING | <ul> <li>Using a two-sided t-test, 90% power and SD =10, 266 patients would be required. Accounting for a 15% drop-out 314 patients are planned to be enrolled.</li> <li>Non-inferiority analysis will be performed after 216 patients, based on OKS at one-year post randomization; MCID is set at 4 points.</li> <li>Using a one-sided t-test, 90% power and SD =10, non-inferiority margin of 4 OKS, 216 patients would be required for the NI analysis.</li> <li>The power calculation is based on reaching sufficient power when a comparison of the study groups is carried out.</li> </ul> |